CLINICAL TRIAL: NCT03826160
Title: Role of Growth Hormone in the Pathogenesis and Treatment of Cardiac Steatosis and Diastolic Dysfunction in HIV
Brief Title: Growth Hormone Dynamics and Cardiac Steatosis in HIV
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Steven K. Grinspoon, MD, Professor of Medicine, Massachusetts General Hospital
Other Study IDs: 2018P001792
Record Dates: First submitted 2019-01-30; First posted 2019-02-01 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Human Immunodeficiency Virus; Lipodystrophy; Cardiac Disease
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Lipodystrophy; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples for subsequent processing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tesamorelin: Individuals who plan to initiate tesamorelin clinically
- No Treatment: Individuals who decline to initiate tesamorelin despite a clinical indication

SUMMARY:
Cardiac steatosis is increased among individuals with HIV, and may predispose to cardiac mechanical dysfunction and subsequent heart failure. The pathogenesis and treatment of cardiac steatosis is not well understood. The investigators have previously shown that perturbed growth hormone (GH) secretion in HIV contributes to ectopic fat accumulation in the viscera and the liver. Moreover, the investigators have found that augmentation of endogenous GH secretion with the FDA-approved medication tesamorelin reduces visceral and hepatic fat. In this longitudinal observational study, the investigators will examine patients with HIV and abdominal fat accumulation who either plan or do not plan to initiate tesamorelin prescribed clinically. The investigators hypothesize that blunted GH secretion in HIV is associated with cardiac steatosis. The investigators also hypothesize that use of tesamorelin for 6 months is associated with a reduction in intramyocardial fat and preserved cardiac function.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, ages 40-70 years
* Documented HIV infection on stable antiretroviral therapy for ≥ 3 months
* Abdominal obesity with waist circumference ≥ 102 cm in men, ≥ 88 cm in women
* Indication for tesamorelin per clinical judgment

Exclusion Criteria:

* CD4 < 100 cells/mm3 or HIV viral load > 400 copies/mL
* Current active AIDS-defining illness
* History or symptoms consistent with heart failure
* Standard contraindications to MRI including severe allergy to gadolinium
* Glomerular filtration rate (eGFR) < 45 mL/min/1.73 m2 within one month of MRI study
* Use of growth hormone-releasing hormone (GHRH) or growth hormone (GH) within the past 6 months
* HbA1c > 7%, chronic insulin use within the past 6 months, and/or change in anti-diabetic agents within the past 3 months
* Change in statin therapy within the past 3 months
* Chronic corticosteroid use except intermittent topic steroid creams or inhalers
* Pregnancy or breastfeeding

Ages: 40 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: HIV patients, age 40-70 years old, with abdominal fat accumulation
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2022-04-19 (Actual); Study Completion 2022-04-19 (Actual)

PRIMARY OUTCOMES:
Intramyocardial lipid content | 6 months
  Measure of fat content within cardiac muscle as assessed by cardiac magnetic resonance spectroscopy (MRS)

SECONDARY OUTCOMES:
Circumferential diastolic strain rate | 6 months
  Measure of diastolic function as assessed by cardiac magnetic resonance imaging (MRI)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Grinspoon, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided